CLINICAL TRIAL: NCT01642732
Title: A Multi-institutional Phase I and Biomarker Study of Everolimus Added to Combined Hormonal and Radiation Therapy for High Risk Prostate Cancer
Brief Title: Study of Everolimus Added to Combined Hormonal and Radiation Therapy for High Risk Prostate Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of accrual and funding expires in June, 2014.
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2011.008; HUM00047650 (Other: Univ Mich Medical School Institutional Review Board (IRBMED))
Record Dates: First submitted 2012-03-24; First posted 2012-07-17 (Estimated); Results first posted 2014-11-20 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Prostate Cancer
Keywords: Prostate; Cancer; Everolimus; Radiation
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — Everolimus; Leuprolide; bicalutamide; Radiation; luprolide acetate gel depot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Everolimus with combined hormonal and radiation therapy (Experimental): Everolimus - there are five dose levels (2.5mg. every 48 hrs.,2.5mg./day, 5mg./day, 7.5mg./day, and 10mg./day) based on the initial expectations of toxicity and the incidence of toxicity of subjects already treated. Subjects will be on one dose level throughout the study. Subjects will receive everolimus starting on study day 1.
  Radiation therapy will start on day 60-70 (44 treatments, at 5 treatments a week for a little longer than 8 weeks).
  Bicalutamide (50 mg. tablets daily) will begin on study day 10-14, approximately 2 months prior to Radiation Therapy.
  Lupron injections will begin on study day 10 to 25, approximately 2 months prior to Radiation Therapy. The typical dose schedule is either one injection (22.5 mg. dose)every 3 months for a total of 8 injections or one injection (30 mg. dose) every 4 months for a total of 6 injections.
  Radiation, bicalutamide, and everolimus will end between study day 120-130. Lupron will end at 24 months on study.
  Interventions: Other: Everolimus, lupron, bicalutamide, and radiation

INTERVENTIONS:
Other: Everolimus, lupron, bicalutamide, and radiation — Everolimus - there are five dose levels (2.5mg. every 48 hrs.,2.5mg./day, 5mg./day, 7.5mg./day, and 10mg./day) based on the initial expectations of toxicity and the incidence of toxicity of subjects already treated. Subjects will be on one dose level throughout the study. Subjects will receive everolimus starting on study day 1.
  Radiation therapy will start on day 60-70 (44 treatments, at 5 treatments a week for a little longer than 8 weeks).
  Bicalutamide (50 mg. tablets daily) will begin on study day 10-14, approximately 2 months prior to Radiation Therapy.
  Lupron injections will begin on study day 15 to 25, approximately 2 months prior to Radiation Therapy. The typical dose schedule is either one injection (22.5 mg. dose)every 3 months for a total of 8 injections or one injection (30 mg. dose) every 4 months for a total of 6 injections.
  Radiation, bicalutamide, and everolimus will end between study day 120-130. Lupron will end at 24 months on study.
  Other Names: afinitor; RAD-001; Casodex; Leuprolide; Eligard

SUMMARY:
The purposes of this study are to:

* Determine the safest and highest dose of the study drug RAD001 (Everolimus) that can be taken in combination with hormonal and radiation therapy in men with high risk prostate cancer.
* Evaluate changes in patient reported quality of life
* Evaluate biomarkers from prostate tumor samples. Biomarkers are various traits which can be used to identify the progress of a disease or condition, which can help researchers determine the effect the study treatment has on the tumor. Biomarkers can also help determine areas for further research.

DETAILED DESCRIPTION:
Prostate cancer is very prevalent with an estimated > 200,000 new cases and > 25,000 deaths attributable to prostate cancer in the United States in 2010. Radiation treatment represents a commonly utilized method to treat prostate cancer with an excellent chance of controlling disease with biochemical control at 5-years in excess of 75% in men with locally confined but intermediate to high-risk disease. However, despite impressive biochemical control, local control remains a problem.

Everolimus is being investigated as an anticancer agent based on its potential to act:

* Directly on the tumor cells by inhibiting tumor cell growth and proliferation
* Indirectly by inhibiting angiogenesis leading to reduced tumor vascularity.

Given the prevalence of PTEN deletion in high-risk prostate cancers as well as the evidence that tumor hypoxia leads to increased risks of failure after treatment with hormonal therapy and radiation, we hypothesis that inhibition of mTOR signaling in both tumor and vascular cells using everolimus concurrent with hormonal and radiation therapy will enhance the efficacy of radiation therapy without an unacceptable risk of toxicity in men with high-risk prostate cancer.

Everolimus has not been approved by the FDA for the treatment of prostate cancer by itself or in combination with radiation and hormonal therapy. It is not known if this combination is safe and effective in prostate cancer. The FDA has allowed their combined use in this clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Participants must be able to care for themselves
* Adequate function
* Adequate kidney function
* Histologically confirmed diagnosis of adenocarcinoma of the prostate with biopsy within 90 days of enrollment
* High-risk prostate cancer
* No distant metastases as evaluated by a bone scan and CT of the pelvis (within 90 days of enrollment)
* Participants must have at least 4 biopsy cores containing prostate cancer with tissue available for histologic analysis
* Signed informed consent

Exclusion Criteria:

* Participants currently receiving anticancer therapies or who have received anticancer therapies within 4 weeks of the start of study drug (including chemotherapy, radiation therapy, antibody based therapy, targeted therapy, etc.)
* Prior pharmacologic androgen ablation for prostate cancer is not allowed including LHRH agonist therapy or oral anti-androgen therapy.

  o Previous use of either finasteride or dutasteride is allowed
* Participants, who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, participants who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia) or participants that may require major surgery during the course of the study
* Any previous therapeutic radiation therapy to the pelvis.
* Known gastrointestinal dysfunction or an inability to take oral medications that would preclude taking an oral medication.
* Prior treatment with any investigational drug within the preceding 4 weeks of registration
* Participants receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent.

  o Topical or inhaled corticosteroids are allowed.
* Participants should not receive immunization with attenuated live vaccines within one week of registration or during study period. Close contact with those who have received attenuated live vaccines should be avoided during treatment with everolimus. Examples of live vaccines include intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella and TY21a typhoid vaccines.
* Other malignancies within the past 3 years except for adequately treated basal or squamous cell carcinomas of the skin.
* Participants who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

  * Symptomatic congestive heart failure of New York heart Association Class III or IV
  * Uncontrolled cardiac arrhythmia
  * The use of anti-arrhythmic medications or implanted pacemakers or defibrillators is allowed and would not exclude a patient from enrollment.
  * Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
  * Severely impaired lung function
  * Uncontrolled diabetes
  * Active (acute or chronic) or uncontrolled severe infections
  * Liver disease such as cirrhosis or severe hepatic impairment
* Uncontrolled diabetes mellitus despite adequate therapy. Patients with a known history of impaired fasting glucose or diabetes mellitus (DM) may be included, however blood glucose and antidiabetic treatment must be monitored closely throughout the trial and adjusted as necessary;
* A detailed assessment of Hepatitis B/C medical history and risk factors must be done at screening for all participants.

  * Participants with previous documented history of Hepatitis B/C infection are excluded from enrollment.
  * Participants with high risk for hepatitis based upon medical history and risk factors must be screened for Hepatitis B and C, and if positive are excluded from enrollment.
* A known history of HIV seropositivity
* Participants with an active, bleeding diathesis
* Male patient whose sexual partner(s) are women of child bearing potential who are not willing to use adequate contraception, during the study and for 8 weeks after the end of treatment
* Participants who have received prior treatment with an mTOR inhibitor (e.g., sirolimus, temsirolimus, everolimus).

  o Sirolimus eluting coronary artery stents are allowed
* Participants with a known hypersensitivity to everolimus or other rapamycins (e.g., sirolimus, temsirolimus) or to its excipients
* Participants unwilling to or unable to comply with the protocol

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-10; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A. Hamstra, M.D., Ph.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (2):
- United States (2):
  - Georgetown University, Washington D.C., District of Columbia
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Everolimus With Combined Hormonal and Radiation Therapy
Started | 1
Completed | 0
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Everolimus With Combined Hormonal and Radiation Therapy
Number analyzed (Participants) | 1
Age, Continuous [Median (Full Range); unit: years] | 54 [54 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events on Oral Everolimus in Combination With Hormonal Ablation and External Beam Radiation
Time Frame: 64 months after beginning everolimus
Population: One patient was enrolled and withdrew from the study prior to treatment. The primary objective was not analyzed.
Arm/Group | Everolimus With Combined Hormonal and Radiation Therapy
Number analyzed (Participants) | 0

2. Secondary Outcome: Difference in Serologic Everolimus and Prostate Biomarker Levels Before and After Treatment With Everolimus
Description: Analysis of pairs of markers will be explored looking for large positive or negative correlations to indicate marker areas for further research.
Time Frame: Prior to treatment and at 14 days
Population: One patient was enrolled and withdrew from the study prior to treatment. The objective was not analyzed.
Arm/Group | Everolimus With Combined Hormonal and Radiation Therapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Only one patient was enrolled and the patient withdrew consent prior to treatment therefore Adverse Events (AEs) and Serious Adverse Events (SAEs) could not be analyzed.
Arm/Group | Everolimus With Combined Hormonal and Radiation Therapy
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Only one patient was enrolled to the trial and consent was withdrawn prior to treatment therefore the primary objective could not be analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes